CLINICAL TRIAL: NCT00807209
Title: A Phase 2 Open-Label, Parallel Group, Randomized, Dose-Finding Study to Assess the Efficacy and Safety of Intercostal SKY0402 in Subjects Undergoing Posterolateral Thoracotomy
Brief Title: Dose Finding Posterolateral Thoracotomy Study
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision unrelated to safety
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SKY0402C211
Record Dates: First submitted 2008-12-09; First posted 2008-12-11 (Estimated); Results first posted 2012-05-15 (Estimated); Last update posted 2012-05-15 (Estimated); Status verified 2011-11

CONDITIONS: Postoperative Pain
Keywords: Pain; postoperative; thoracotomy
MeSH Terms: conditions — Pain, Postoperative; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- High Dose SKY0402 (Experimental)
  Interventions: Drug: High Dose SKY0402; Drug: Fentanyl via PCA; Drug: Bupivacaine via epidural
- Standard of Care (Active Comparator)
  Interventions: Drug: Placebo; Drug: Fentanyl via PCA; Drug: Bupivacaine via epidural
- Low Dose SKY0402 (Experimental)
  Interventions: Drug: Low Dose SKY0402; Drug: Fentanyl via PCA; Drug: Bupivacaine via epidural

INTERVENTIONS:
Drug: Low Dose SKY0402 — Bupivacaine, 15 mg/mL via epidural PLUS single total administration of 75mg SKY0402 (25 mg to each of three segments) in 4 mL volume each for a total of 12 mL via nerve block (intercostal)
  Arms: Low Dose SKY0402
Drug: High Dose SKY0402 — Bupivacaine, 15 mg/mL via epidural PLUS single total administration of 150 mg (50 mg to each of three segments) in 4 mL volume each for a total of 12 mL via nerve block (intercostal)
  Arms: High Dose SKY0402
Drug: Placebo — Bupivacaine, 15 mg/mL per epidural PLUS administration of 4 mL Placebo to each of three nerves for a total of 12 mL (intercostal)
  Arms: Standard of Care
Drug: Fentanyl via PCA — Fentanyl via PCA
Drug: Bupivacaine via epidural — Bupivacaine via epidural

SUMMARY:
To review safety and effectiveness of two doses compared to current standard of care.

DETAILED DESCRIPTION:
Evaluate the efficacy of intercostal nerve block using SKY0402 compared to epidural bupivacaine HCl in subjects undergoing posterolateral thoracotomy. The primary outcome metric for this will be the amount of rescue PCA fentanyl administered for breakthrough pain during the first 72 hours.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥ 18 years of age at the Screening Visit.
* Scheduled to undergo a thoracotomy of at least 3 inches of intercostal incisional length or requiring insertion of an inter-rib spreader/retractor for a primary thoracic non-infectious indication under general anesthesia.
* Able and willing to receive an epidural catheter for the treatment of postoperative pain.
* American Society of Anesthesiology (ASA) Physical Class 1-4.
* Able and willing to comply with all study visits and procedures.
* Able to speak, read, and understand the language of the ICF, study questionnaires, and other instruments used for collecting subject-reported outcomes, in order to enable accurate and appropriate responses to pain scales and other required study assessments.
* Willing and capable of providing written informed consent.

Exclusion Criteria:

* Known metastatic disease of any type.
* Known pulmonary infectious disease.
* Pregnancy, nursing, or planning to become pregnant during the study or within one month after study drug administration.
* Use of any of the following medications within the times specified before surgery:

  1. Long-acting opioids within 3 days.
  2. Any opioid medication within 24 hours.
* Concurrent painful physical condition or concurrent surgery that may require analgesic treatment in the postoperative period for pain that is not strictly related to the surgical site being administered study drug (e.g., significant pain from other joints, chronic neuropathic pain, concurrent abdominal surgery, etc.), which have the potential to confound the postoperative study assessments.
* Body weight less than 50 kilograms (110 pounds).
* History of hypersensitivity or idiosyncratic reaction to amide-type local anesthetics, opioid medication, epinephrine, or sulfites.
* Contraindication to epinephrine, such as concurrent administration of ergot-type drugs, monoamine oxidase (MAO) inhibitors or antidepressants of tryptoline or imipramine types, conditions where the production or exacerbation of tachycardia could prove fatal (e.g., poorly controlled thyrotoxicosis or severe heart disease), or any other pathological conditions that might be aggravated by the effects of epinephrine.
* Administration of an investigational product within 30 days or 5 elimination half-lives of such investigational product, whichever is longer, prior to study drug administration, or planned administration of another investigational product or procedure during the subject's participation in this study.
* History of, suspected, or known addiction to or abuse of illicit drug(s), prescription medicine(s), or alcohol within the past 2 years.
* Uncontrolled anxiety, schizophrenia, or other psychiatric disorder that, in the opinion of the Investigator, may interfere with study assessments or compliance with the protocol.
* Significant medical conditions or laboratory results that, in the opinion of the Investigator, indicate an increased vulnerability to study drugs and procedures, and expose the subject to an unreasonable risk as a result of participating in this clinical trial, such as: debilitating diseases, acute illnesses, hypotension, partial or complete conduction block, impaired cardiac function, untreated hypertension, advanced arteriosclerotic heart disease, cerebral vascular insufficiency, pre-existing abnormal neurological or neuromuscular disease (e.g., epilepsy, myasthenia gravis), advanced liver disease, sever renal impairment, advanced diabetes, co-morbid conditions associated with an immunocompromised status, such as blood dyscrasias, HIV/AIDS, or recent chemotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2008-12; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kay Warnott, RN, ACN-P, Study Director — Pacira Pharmaceuticals, Inc
Locations (5):
- United States (5):
  - Lotus Clinical Research, Pasadena, California
  - Florida Hospital, Orlando, Florida
  - Memorial Hermann - Memorial City Medical Center, Houston, Texas
  - Houston NW Medical Center, Houston, Texas
  - Multicare Health System, Tacoma, Washington

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | High Dose SKY0402 | Standard of Care | Low Dose SKY0402
Started | 1 | 1 | 1
Completed | 1 | 1 | 1
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Dose SKY0402 | Standard of Care | Low Dose SKY0402 | Total
Number analyzed (Participants) | 1 | 1 | 1 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 1 | 1
  >=65 years | 1 | 1 | 0 | 2
Age Continuous [Mean (Standard Deviation); unit: years] | 81 (0) | 75 (0) | 64 (0) | 73.3 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1 | 2
  Male | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Amount of Rescue PCA Fentanyl Administered for Breakthrough Pain During the First 72 Hours.
Description: The primary outcome metric was to be the amount of rescue epidural fentanyl administered for breakthrough pain during the first 72 hours postoperatively. Patient-controlled analgesia (PCA) fentanyl intake was to be summarized for each treatment group as time to first use of rescue PCA fentanyl, amount of PCA fentanyl administered over 72 hours, and total amount of PCA fentanyl administered through a number of time intervals. However, efficacy analyses were not performed because the study was terminated early after only three subjects were enrolled.
Time Frame: 72 hours
Measure: Number; unit: micrograms
Groups:
- High Dose SKY0402; Low Dose SKY0402: Single dose of study drug divided equally into three 4 mL doses and delivered to each of three nerve segments following posterolateral thoracotomy
- Standard of Care: Bupivacaine HCl solution (1.25 mg/mL) and epinephrine (5 mcg/mL) administered via an epidural catheter at a concentration of 0.125% (1.25 mg/mL) at a rate of 8 cc per hour
Arm/Group | High Dose SKY0402 | Standard of Care | Low Dose SKY0402
Number analyzed (Participants) | 0 | 1 | 1
micrograms |  | 0 | 0

ADVERSE EVENTS:
Arm/Group | High Dose SKY0402 | Standard of Care | Low Dose SKY0402
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 1/1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | High Dose SKY0402 (N=1) | Standard of Care (N=1) | Low Dose SKY0402 (N=1)
Gas (Gastrointestinal disorders) | 0 | 1 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 0
Swollen Ankle (Injury, poisoning and procedural complications) | 0 | 1 | 0
Difficulty breathing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Blood in nasal mucus (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
The study was terminated early due to Sponsor's decision, unrelated to safety. As there was only one patient in each group, no efficacy analyses were performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No